CLINICAL TRIAL: NCT03597906
Title: Comparison of the Outcome of Topography Modified Refraction Correction to Standard Clinical Refraction Correction in Myopic Astigmatic Topography-guided LASIK
Brief Title: Topography Guided LASIK by Different Protocols for Treatment of Astigmatism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Fayrouz Aboalazayem, the principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: N-18-2018
Record Dates: First submitted 2018-06-21; First posted 2018-07-24 (Actual); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Refractive Surgery
Keywords: Topography guided ablation; Astigmatism; LASIK
MeSH Terms: conditions — Astigmatism

STUDY DESIGN:
Intervention Model Description: A prospective, randomized and comparative interventional study
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group A: Manifest (Experimental): 20 eyes will be treated using Contoura, topography guided ablation vision with the standard manifest refraction.
  Interventions: Procedure: topography guided ablation; Procedure: manifest refraction
- Group B: partial TMR (Experimental): 20 eyes will be treated with Contoura vision, topography guided ablation using the topographic astigmatic power and axis and without change in the spherical power (using the same spherical power as the manifest refraction).
  Interventions: Procedure: topography guided ablation; Procedure: partial topography modified refraction
- Group C: Full TMR (Experimental): 20 eyes will be treated with Contoura vision, topography guided ablation using the topographic astigmatic power and axis and modifying the spherical power to obtain the same spherical equivalent as the manifest refraction. This is done by subtracting half of the difference between topographic astigmatic power and the manifest astigmatic power from the spherical power (topography-modified treatment refraction).
  Interventions: Procedure: topography guided ablation; Procedure: full topography modified refraction

INTERVENTIONS:
Procedure: topography guided ablation — using the data obtained from the topolyzer for correction of refractive errors specially astigmatism we use 3 different treatment protocols
Procedure: manifest refraction — using for ablation the exact manifest refraction
  Arms: Group A: Manifest
Procedure: full topography modified refraction — full topography modified refraction means changing both sphere and cylinder power in the ablation profile
  Arms: Group C: Full TMR
Procedure: partial topography modified refraction — partial topography modified refraction means changing only cylinder power and axis in the ablation profile
  Arms: Group B: partial TMR

SUMMARY:
Background and Rationale:

LASIK has been among the highest satisfaction rates of surgical procedures, ranging from 82%-98%. Different ablation profiles have been developed over the years. The purpose of this study is to validate this novel measurement by comparing the visual outcomes when the TMR is used in myopic astigmatic LASIK to using the standard manifest refraction or the Topolyzer measurements alone.

Objectives :

To evaluate the safety, efficacy and predictability of topography-guided myopic LASIK with three different refraction treatment strategies.

DETAILED DESCRIPTION:
Candidates for refractive surgery above 18 years with myopic astigmatism and no previous ocular surgery.

Sample size 60 eyes. surgery:

* 60 eyes of myopic topography-guided LASIK procedures with the same refractive platform (FS200 femtosecond to create a flap between90: 110 μm with diameter 8:9 mm and EX500 excimer lasers) will be randomized for treatment as follows:
* Group A: 20 eyes will be treated using Contoura vision with the standard manifest refraction.
* Group B: 20 eyes will be treated with Contoura vision using the topographic astigmatic power and axis and without change in the spherical power (using the same spherical power as the manifest refraction).
* Group C [TMR]: 20 eyes will be treated with Contoura vision using the topographic astigmatic power and axis and modifying the spherical power to obtain the same spherical equivalent as the manifest refraction. This is done by subtracting half of the difference between topographic astigmatic power and the manifest astigmatic power from the spherical power (topography-modified treatment refraction).
* The standard postoperative treatment is combined steroids and antibiotics eye drops 5 times daily for one week ,then three times daily for three days and lubricant eye drops 5 times daily for six months.

Postoperatively, the patients will be examined at 1 week, 1 month and 3 months. All postoperative follow-up visits included measurement of UDVA, CDVA (if indicated) and refraction, besides full ophthalmological examination and performing pentacam and topolyzer after 3 months

ELIGIBILITY:
Inclusion Criteria:

* Stable refractive error: Myopic astigmatism ≥ -1.5 D
* Valid Topolyzer maps (at least four out of eight right maps with green analyzed area and the registration box is green).

Exclusion Criteria:

1. Estimated postoperative residual stromal bed thickness of less than 300µm.
2. Glaucomatous patients.
3. Patients with keratoconus.
4. Patients with pervious refractive surgery.
5. History of previous ocular trauma or surgery.
6. History of recent herpetic ulcer or viral keratitis.
7. Basement membrane disease, history of recurrent corneal erosions.
8. Sicca syndrome, dry eye.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-08-15 (Actual); Primary Completion 2019-11-15 (Actual); Study Completion 2020-01-20 (Actual)

PRIMARY OUTCOMES:
post operative residual astigmatism | 3 months
  measuring the post operative residual astigmatism and comparison between the 3 group to reach to the most accurate protocol.

SECONDARY OUTCOMES:
measurement of the postoperative unaided visual acuity | 3 months
  measurement of the postoperative unaided visual acuity and comparison between the 3 group to reach to the most accurate protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Mohmed Hosny, MD, Study Director — Cairo University
Locations (1):
- Kasr Alainy, Cairo, Egypt